CLINICAL TRIAL: NCT05933772
Title: Performance Evaluation of Two Silicone Hydrogel Toric Lens Designs in Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-149
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, Then Lens B (Experimental): Participants will wear Lens A for one month and then crossover to Lens B for one month.
  Interventions: Device: Lens A (comfilcon A toric lens); Device: Lens B (lehfilcon A toric lens)
- Lens B, Then Lens A (Experimental): Participants will wear Lens B for one month and then crossover to Lens A for one month.
  Interventions: Device: Lens A (comfilcon A toric lens); Device: Lens B (lehfilcon A toric lens)

INTERVENTIONS:
Device: Lens A (comfilcon A toric lens) — One month wear
Device: Lens B (lehfilcon A toric lens) — One month wear

SUMMARY:
The objective of the study was to compare the clinical performance of two monthly toric silicone hydrogel contact lenses in habitual wearers, when worn for 1-month each.

DETAILED DESCRIPTION:
This study was a prospective, bilateral eye, subjected-masked, randomized, 1-month cross-over, daily-wear design involving two different silicone hydrogel toric lens types. Each lens type will be worn bilaterally for approximately one month.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 39 years of age (inclusive) and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self-reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 6 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears of toric soft contact lenses binocularly.

   1. No more than 1/3 of the participants should be wearing daily disposable soft toric lenses;
   2. the remaining 2/3+ of the participants must be planned frequent replacement soft toric lens wearers as follows:

      * i. TOTAL30 for Astigmatism: maximum of 3 (∼10%) (no target percentage)
      * ii. Biofinity toric: maximum of 13 (∼40%) (PLUS a target of minimum 10 (∼30%))
      * iii. Air Optix for Astigmatism (inclusive of +Hydraglyde): maximum of 10 (∼30%) (PLUS a target of minimum 7 (∼20%))
      * iv. ULTRA for Astigmatism: maximum of 5 (∼15%) (no target percentage)
      * v. Acuvue Vita for Astigmatism: maximum of 3 (∼10%) (no target percentage)
      * vi. Acuvue Oasys for Astigmatism: maximum of 10 (∼30%) (no target percentage)
      * vii. Other brands of frequent replacement: maximum of 7 (∼20%) (no target percentage)
7. Has refractive astigmatism of at least -0.75DC but no more than -2.75DC in each eye that is correctable with a soft toric lens with a cylinder power of no greater than -2.25DC;
8. Is ammetropic and requires a spectacle spherical component of +8.00 to -10.00D inclusively;
9. Can be fit and achieve binocular distance vision of at least 20/32 Snellen with the available lens parameters

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active ocular disease and/or infection that contraindicates contact lens wear;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sacco, Principal Investigator — Sacco Eye Group; David Wilkinson, Principal Investigator — Spadina Optometry; Fiona Soong, Principal Investigator — Eyes on Sheppard Clinic; Katherine Bickle, Principal Investigator — ProCare Vision Center; Shane R. Kannarr, Principal Investigator — Kannarr Eye Care
Locations (5):
- United States (3):
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Center, Granville, Ohio
- Canada (2):
  - Eyes on Sheppard Clinic, Toronto, Ontario
  - Spadina Optometry, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 50 participants enrolled and 1 was discontinued due to lost to follow-up prior to the first lens dispense.
Period: First Intervention, 1 Month
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0
Period: Second Intervention, 1 Month
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis Population
Groups:
- Analysis Population: All participants who completed study. (Total Study Population n=49)
Arm/Group | Analysis Population
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling on Removal
Description: Lens Handling on Removal, using a 0-100 scale (0= very difficult, 100=very easy).
Time Frame: At the end of one month of wear
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Participants that received Lens A during either the first or second period of the study.
- Lens B: Participants that received Lens B during either the first or second period of the study.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 49 | 49
units on a scale | 89 (17) | 91 (14)

2. Secondary Outcome: Distance Visual Acuity
Description: Distance Visual Acuity, using Snellen converted to logMAR.
Time Frame: At the end of one month of wear
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 49 | 49
logMAR | -0.06 (0.06) | -0.06 (0.06)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 months.
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 5/49 | 4/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (N=49) | Lens B (N=49)
Inflammated skin due to eye make-up spread in eye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Red Eye (No Discomfort) (Eye disorders) | 1 (1) | 0 (0)
Botox Injection (General disorders) | 1 (1) | 0 (0)
Gum Graft Surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnolence (General disorders) | 0 (0) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stuffy nose and sneezing (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT05933772/Prot_SAP_000.pdf